CLINICAL TRIAL: NCT00706264
Title: Randomized Controlled Trial: Prevention of Preterm Birth Using Cervical Pessary in Pregnant Women With Short Cervix (PECEP)
Brief Title: Prevention of Preterm Birth Using Cervical Pessary in Pregnant Women With Short Cervix
Acronym: PECEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maternal-Infantil Vall d´Hebron Hospital (Other)
Collaborators: Hospital Universitario de Canarias (Other); Hospital Son Llatzer (Other); Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Maria Goya, MD, PhD, PhD, Maternal-Infantil Vall d´Hebron Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PECEP-TRIAL
Record Dates: First submitted 2008-06-24; First posted 2008-06-27 (Estimated); Results first posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Preterm Birth
Keywords: Short cervix; preterm birth; arabin pessary
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Expectant management
- 2 (Experimental): Placement of arabin pessary since 23 weeks until 37 weeks
  Interventions: Device: Silicon ring (Arabin Pessary)

INTERVENTIONS:
Device: Silicon ring (Arabin Pessary) — Placement of a silicon pessary in the vagina, around the cervix.
  Other Names: Vaginal pessaries CE 0482 MED / CERT ISO 9003 /EN 46003
  Arms: 2

SUMMARY:
Placement of a vaginal pessary reduces significantly the rate of spontaneous preterm birth in pregnant women with short cervical length at 18-22 weeks scan.

DETAILED DESCRIPTION:
This trial includes pregnant women undergoing routine ultrasound examination at 18.0 to 22.6 weeks of gestation.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Minimal age of 18 years

Exclusion Criteria:

* Major fetal abnormalities (requiring surgery or leading to infant death or severe handicap)
* SROM at the time of randomization
* Cervical cerclage in situ
* Active vaginal bleeding
* Previous cone biopsy or cerclage
* Major uterine structural anomalies
* Placenta previa

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 385 (Actual)
Dates: Start 2007-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ELENA CARRERAS, PhD, Study Director — Maternal-Infantil Vall d´Hebron Hospital
Locations (6):
- Spain (6):
  - Hospital Materno-Infantil de Canarias, Las Palmas de Gran Canaria, Gran Canaria
  - Hospital Son Llàtzer, Palma de Mallorca, Mallorca
  - Hospital de Reus, Reus, Tarragona
  - Hospital Vall d´Hebron, Barcelona
  - Institut Universitary Dexeus, Barcelona
  - Hospital de Fuenlabrada, Madrid

REFERENCES:
- [Derived] Goya M, Pratcorona L, Merced C, Rodo C, Valle L, Romero A, Juan M, Rodriguez A, Munoz B, Santacruz B, Bello-Munoz JC, Llurba E, Higueras T, Cabero L, Carreras E; Pesario Cervical para Evitar Prematuridad (PECEP) Trial Group. Cervical pessary in pregnant women with a short cervix (PECEP): an open-label randomised controlled trial. Lancet. 2012 May 12;379(9828):1800-6. doi: 10.1016/S0140-6736(12)60030-0. Epub 2012 Apr 3. PMID 22475493

RESULTS

PARTICIPANT FLOW:
Recruitment Details: You are right that our fi rst planned sample size was 2780 patients. However, after the first interim analysis, and in accordance with the advice of our Data Monitoring Committee, the protocol was amended to reach the new and fi nal sample size.
Groups:
- Expectant Management: Expectant management: Current conventional management.
- Placement of Arabin Pessary Since 23 Weeks Until 37 Weeks: Placement of arabin pessary since 23 weeks until 37 weeks
  Silicon ring (Arabin Pessary): Placement of a silicon pessary in the vagina, around the cervix.
Period: Overall Study
Arm/Group | Expectant Management | Placement of Arabin Pessary Since 23 Weeks Until 37 Weeks
Started | 193 | 192
Completed | 190 | 190
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Expectant Management: Both groups were seen by the clinical team of the trial at each centre every month until delivery. Transabdominal ultrasonography was done for fetal biometries and wellbeing, clinical questionnaire was administered for confi rmation of correct device placement in the pessary group (fi gure 2), vaginal swab was taken for study of bacteriological infection, and transvaginal ultra sonography was done to measure cervical length (fi gure 3)
- Placement of Arabin Pessary Since 23 Weeks Until 37 Weeks: The pessary was removed during the 37th week of gestation. Indications for pessary removal before this time were active vaginal bleeding, risk of preterm labour with persistent contractions despite tocolysis, or severe patient discomfort.
- Total: Total of all reporting groups
Arm/Group | Expectant Management | Placement of Arabin Pessary Since 23 Weeks Until 37 Weeks | Total
Number analyzed (Participants) | 190 | 190 | 380
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 190 | 190 | 380
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (5.4) | 30.3 (5.1) | 30.1 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 190 | 380
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56 | 58 | 114
  Not Hispanic or Latino | 134 | 132 | 266
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 190 | 190 | 380

OUTCOME MEASURES:

1. Primary Outcome: Spontaneous Delivery Before 34 Completed Weeks
Description: Number of spontaneous preterm births before 34 weeks occurred in each group.
Time Frame: Between 24 and 34 weeks
Measure: Count of Participants; unit: Participants
Groups:
- No Intervention: No Pessary: No pessary will be used. Subjects will receive standard obstetrical care and management.
- Experimental: Pessary: Use of Arabin pessary. Pessary placed around the cervix between 20 and 23 weeks gestation, and will be removed during the 37th week of pregnancy.
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 190 | 190
Participants | 51 | 12

2. Secondary Outcome: Birthweight Less Than 1500 g
Description: Number of newborns whose birthweight is less than 1500 grams
Time Frame: Time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 190 | 190
Participants | 26 | 9

3. Secondary Outcome: Birthweight Less Than 2500 g
Description: Number of newborns whose birthweight is less than 2500 grams
Time Frame: Time of delivery
Measure: Count of Participants; unit: Participants
Groups:
- Expectant Management: Expectant management: usual management
- Placement of Arabin Pessary Since 23 Weeks Until 37 Weeks: Silicon ring (Arabin Pessary): Placement of a silicon pessary in the vagina, around the cervix.
Arm/Group | Expectant Management | Placement of Arabin Pessary Since 23 Weeks Until 37 Weeks
Number analyzed (Participants) | 190 | 190
Participants | 56 | 17

4. Secondary Outcome: Intrauterine Fetal Demise
Description: The number of fetal deaths in the pessary group was compared to those in the no pessary group
Time Frame: Pregnancy
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 190 | 190
Participants | 0 | 0

5. Secondary Outcome: Neonatal Death
Description: The number of neonatal deaths in the pessary group was compared to those in the no pessary group
Time Frame: Between birth and 28 days of age
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 190 | 190
Participants | 1 | 0

6. Secondary Outcome: Intraventricular Haemorrhage
Description: The number of neonatal intraventricular haemorrhage in the pessary group was compared to those in the no pessary group
Time Frame: Between birth and 28 days of age
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 190 | 190
Participants | 2 | 0

7. Secondary Outcome: Respiratory Distress Syndrome
Description: The number of neonatal Respiratory distress syndrome in the pessary group was compared to those in the no pessary group
Time Frame: Between birth and 28 days of age
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 190 | 190
Participants | 23 | 5

8. Secondary Outcome: Retinopathy of Prematurity
Description: The number of neonatal retinopathy in the pessary group was compared to those in the no pessary group
Time Frame: Between birth and 28 days of age
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 190 | 190
Participants | 2 | 0

9. Secondary Outcome: Necrotising Enterocolitis
Description: The number of neonatal necrotising enterocolitis in the pessary group was compared to those in the no pessary group
Time Frame: Between birth and 28 days of age
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 190 | 190
Participants | 2 | 0

10. Secondary Outcome: Treatment for Sepsis
Description: The number of neonatal cases of treatment needed for sepsis in the pessary group was compared to those in the no pessary group
Time Frame: Between birth and 28 days of age
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 190 | 190
Participants | 12 | 3

11. Secondary Outcome: Composite Adverse Outcomes
Description: The number of neonatal cases with composite adverse outcomes in the pessary group was compared to those in the no pessary group
Time Frame: Between birth and 28 days of age
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 190 | 190
Participants | 30 | 5

12. Secondary Outcome: Spontaneous Delivery Before 28 Completed Weeks
Description: Number of preterm births before 28 weeks occurred in each group.
Time Frame: Between 24 and 28 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 190 | 190
Participants | 16 | 4

13. Secondary Outcome: Any Delivery Before 34 Completed Weeks
Description: Number of all preterm births before 34 weeks occurred in each group.
Time Frame: Between 24 and 34 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 190 | 190
Participants | 53 | 14

14. Secondary Outcome: Spontaneous Delivery Before 37 Completed Weeks
Description: Number of preterm births before 37 weeks occurred in each group.
Time Frame: Between 24 and 37 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 190 | 190
Participants | 113 | 41

15. Secondary Outcome: Gestational Age at Delivery
Description: Number of weeks of gestation completed by time of delivery
Time Frame: At time of birth
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 190 | 190
weeks | 34.9 (4.0) | 37.7 (2.0)

16. Secondary Outcome: Use of Tocolysis
Description: Number of participants required use of tocolytic medication
Time Frame: participants will be followed for the duration of pregnancy, up to nine months
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 190 | 190
Participants | 101 | 64

17. Secondary Outcome: Use of Antenatal Steroids
Description: Number of participants that received betamethasone to reduce morbidity of expected preterm delivery
Time Frame: participants will be followed for the duration of pregnancy, up to nine months
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 190 | 190
Participants | 121 | 80

18. Secondary Outcome: Chorioamnionitis
Description: Number of participants that showed intrauterine infection diagnosed by maternal tachycardia, fever, uterine tenderness, purulent or abnormal cervical discharge, fetal tachycardia.
Time Frame: participants will be followed for the duration of pregnancy, up to nine months
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 190 | 190
Participants | 6 | 5

19. Secondary Outcome: Vaginal Bleeding
Description: Number of participants who experienced bleeding from lower genital tract during antepartum period
Time Frame: participants will be followed for the duration of pregnancy, up to nine months
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 190 | 190
Participants | 9 | 7

20. Secondary Outcome: Preterm Premature Rupture of Membranes
Description: Number of participants who experienced rupture of membranes as diagnosed by speculum exam showing pooling, ferning, positive nitrazine test, positive amnisure test.
Time Frame: participants will be followed for the duration of pregnancy, up to nine months
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 190 | 190
Participants | 17 | 3

21. Secondary Outcome: Cesarean Delivery
Description: Number of participants that underwent cesarean delivery
Time Frame: At time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 190 | 190
Participants | 40 | 41

22. Secondary Outcome: Vaginal Discharge
Description: Number of participants who experienced an increased vaginal discharge.
Time Frame: participants will be followed for the duration of pregnancy, up to nine months
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 190 | 190
Participants | 87 | 190

23. Secondary Outcome: Pessary Repositioning Without Removal
Description: Number of participants who required pessary repositioning without removal. This outcome measure only applied to the Experimental (Pessary Arm) and no data were collected from participants in the No Intervention _(No Pessary Arm).
Time Frame: participants will be followed for the duration of pregnancy, up to nine months
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 0 | 190
Participants | 0 | 27

24. Secondary Outcome: Pessary Withdrawal
Description: Number of participants who experience pessary withdrawal. This outcome measure only applied to the Experimental (Pessary Arm) and no data were collected from participants in the No Intervention _(No Pessary Arm).
Time Frame: participants will be followed for the duration of pregnancy, up to nine months
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention: No Pessary | Experimental: Pessary
Number analyzed (Participants) | 0 | 190
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Starting at 24 weeks until 28 days after birth
Arm/Group | Expectant Management | Placement of Arabin Pessary Since 23 Weeks Until 37 Weeks
All-Cause Mortality (participants affected / at risk) | 0/190 | 0/190
Serious Adverse Events (participants affected / at risk) | 0/190 | 0/190
Other Adverse Events (participants affected / at risk) | 0/190 | 0/190

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No